CLINICAL TRIAL: NCT05228249
Title: Loncastuximab Tesirine in Combination With BEAM (Carmustine, Etoposide, Ara-C, Melphalan) Conditioning Regimen Prior to Autologous Stem Cell Transplant (ASCT) and for Maintenance Therapy in Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Loncastuximab Tesirine in Combination With Chemotherapy Prior to Stem Cell Transplant for the Treatment of Recurrent or Refractory Diffuse Large B-Cell Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left institution and funding sponsor closed study. Study did not open to accrual, and no participants were enrolled.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: ADC Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1121551; NCI-2021-14126 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10881 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Recurrent Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Refractory Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Refractory Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Stem Cell Transplantation; Carmustine; Cytarabine; Etoposide; loncastuximab tesirine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (loncastuximab tesirine, BEAM chemotherapy) (Experimental): PART I (CONDITIONING): Patients receive loncastuximab tesirine IV on day -7, carmustine IV over 2 hours on day -7, etoposide IV over 1-2 hours BID days -6, -5, -4, and -3, cytarabine IV over 1 hour BID on days -6, -5, -4, and -3, and melphalan IV over 15-20 minutes on day -2. Patients undergo peripheral blood ASCT per standard practice on day 0.
  PART II (MAINTENANCE): Beginning 30-90 days after ASCT, patients receive loncastuximab tesirine IV Q3V for up to 9 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Drug: Cytarabine; Drug: Etoposide; Biological: Loncastuximab Tesirine; Drug: Melphalan

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo peripheral blood ASCT
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Biological: Loncastuximab Tesirine — Given IV
  Other Names: ADC ADCT-402; ADCT-402; Anti-CD19 PBD-conjugate ADCT-402; Loncastuximab Tesirine-lpyl; Zynlonta
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813

SUMMARY:
This phase I trial studies the side effects and best dose of loncastuximab tesirine in combination with carmustine, etoposide, cytarabine, and melphalan (BEAM) chemotherapy regimen in treating patients with diffuse large B-cell lymphoma that has come back (recurrent) or has not responded to treatment (refractory). Loncastuximab tesirine is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Chemotherapy drugs, such as carmustine, etoposide, cytarabine, and melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy with loncastuximab tesirine may kill more cancer cells.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of loncastuximab tesirine.

PART I (CONDITIONING): Patients receive loncastuximab tesirine intravenously (IV) on day -7, carmustine IV over 2 hours on day -7, etoposide IV over 1-2 hours twice daily (BID) days -6, -5, -4, and -3, cytarabine IV over 1 hour BID on days -6, -5, -4, and -3, and melphalan IV over 15-20 minutes on day -2. Patients undergo peripheral blood ASCT per standard practice on day 0.

PART II (MAINTENANCE): Beginning 30-90 days after ASCT, patients receive loncastuximab tesirine IV once every 3 weeks (Q3W) for up to 9 cycles in the absence of disease progression or unacceptable toxicity.

After completion of the study treatment, patients are followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PART 1: Subjects must have a histologically confirmed diagnosis of diffuse large B-cell lymphoma including diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B-cell lymphoma, high grade B-cell lymphoma (with MYC and BCL-2 and/or BCL-6 gene rearrangement), and DLBCL arising from follicular lymphoma
* PART 1: Subjects must be eligible for high-dose therapy (BEAM conditioning chemotherapy) and autologous stem cell transplant, as determined by transplant center
* PART 1: Subjects must have chemosensitive disease as defined radiographically (positron emission tomography [PET]/computed tomography [CT] and/or diagnostic CT) by at least a partial response (PR) to their last cycle of salvage therapy, within 60 days of enrollment
* PART 1: Subjects must be >= 18 years of age
* PART 1: Eastern Cooperative Oncology Group (ECOG) score =< 2 or Karnofsky score >= 60%
* PART 1: Creatinine clearance (CrCl) > 40 mL/min by Cockcroft-Gault formula or serum creatinine =< 2.0 mg/dL
* PART 1: Total bilirubin =< 1.5 x the upper limit of normal (ULN) unless isolated hyperbilirubinemia attributed to Gilbert's syndrome; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN
* PART 1: Adequate pulmonary function, defined as lung carbon monoxide diffusing capability test (DLCO) (corrected or uncorrected for hemoglobin per institutional standards), forced expiratory volume in 1 (FEV1), forced vital capacity (FVC) >= 50% of predicted
* PART 1: Cardiac: Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) of >= 50%. Patients 60 years or older must have an LVEF at rest >= 40%, as measured by echocardiogram or radionuclide ventriculogram scan (MUGA)
* PART 1: Hematologic: Prothrombin time (PT)/international normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time PTT) (activated partial thromboplastin time [aPTT]) < 1.5 x ULN, absolute neutrophil count (ANC) >= 1000/mL, platelet >= 75,000/uL
* PART 1: Women of childbearing potential (WOCBP), defined as those who have not been surgically sterilized or who have not been free of menses for at least 1 year, must have a negative serum pregnancy test within 7 days of and prior to initiating loncastuximab tesirine in combination with BEAM conditioning

  * Fertile male and WOCBP subjects must be willing to use highly effective contraceptive methods before, during, and for at least 6 months after ASCT or 9 months after the last administration of loncastuximab tesirine for women, 6 months after the last administration of loncastuximab tesirine for men, whichever is longer
* PART 1: Ability to provide informed consent
* PART 2: Eligible disease status. Following ASCT (within day +30 to +90), subjects must have achieved radiographic partial response (PR) or complete response (CR) via PET/CT and/or diagnostic CT
* PART 2: Targeted radiation therapy following ASCT is allowed but must be completed >= 2 weeks prior to starting maintenance therapy
* PART 2: Performance status ECOG 0-2 and/or Karnofsky >= 60
* PART 2: CrCl > 40 mL/min by Cockcroft-Gault formula or serum creatinine =< 2.0 mg/dL
* PART 2: Total bilirubin =< 1.5 x the upper limit of normal (ULN) unless isolated hyperbilirubinemia attributed to Gilbert's syndrome; AST and ALT =< 3 x ULN
* PART 2: PT/INR < 1.5 x ULN and PTT (aPTT) < 1.5 x ULN, ANC >= 1000/mL, platelet >= 75,000/mL
* PART 2: Pregnancy and the need for contraception. Negative serum pregnancy test within 7 days of initiating loncastuximab tesirine as maintenance therapy for women of childbearing potential (WOCBP), defined as those who have not been surgically sterilized or who have not been free of menses for at least 1 year

  * Fertile male and WOCBP patients must be willing to use highly effective contraceptive methods before, during, and for at least 6 months after ASCT or 16 weeks after the last administration of loncastuximab tesirine, whichever is longer

Exclusion Criteria:

* PART 1: Receiving other investigational agents
* PART 1: History of central nervous system (CNS) involvement by lymphoma
* PART 1: If a history of receiving a CD19 targeting agent (e.g., CD19 directed CAR T-cell Kymriah, Yescarta, Breyanzi, CD19 antibody Monjuvi), must have pathologic evidence for CD19 expression after receiving CD19 targeting agent
* PART 1: History of immunogenicity or hypersensitivity to a CD19 antibody
* PART 1: Uncontrolled bacterial, viral or fungal infection (currently taking medication and with progression or no clinical improvement); symptomatic congestive heart failure unresponsive to treatment, unstable angina pectoris, symptomatic cardiac arrhythmia not including premature ventricular contractions (PVC); or psychiatric illness/social situations that would limit compliance with study requirements
* PART 1: Active autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, Sjogren's syndrome, autoimmune vasculitis [e.g., granulomatosis with polyangiitis]); motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis); other central nervous system (CNS) autoimmune disease (e.g., poliomyelitis, multiple sclerosis)
* PART 1: Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath)
* PART 1: Known seropositivity for human immunodeficiency virus (HIV), known history of hepatitis B or hepatitis C
* PART 1: Active second primary malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that the investigator(s) agreed and had documented that it was not exclusionary
* PART 1: Any other significant medical illness, abnormality, or condition that could, in the investigator(s)' judgment, make the patient inappropriate for study participation or could put the patient at risk
* PART 1: Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on bone marrow biopsy prior to initiation of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (Part 1) | Up to 30 days
  Will be descriptive based on the appropriate analysis set and may include summary statistics such as means/median, standard deviations, range for continuous variables, and count/percentage for categorical variables, if applicable.
Incidence of toxicity requiring dose delay or modification (Part 2) | Up to 30 days
  Will be descriptive based on the appropriate analysis set and may include summary statistics such as means/median, standard deviations, range for continuous variables, and count/percentage for categorical variables, if applicable.

SECONDARY OUTCOMES:
Progression-free survival | Time from receiving loncastuximab tesirine to the first observation of disease progression or death from any cause, whichever occurs first, assessed at 2 years post-autologous stem cell transplantation (ASCT)
  Kaplan-Meier curves and median time-to-event estimation with 95% confidence intervals will be presented for time to-event endpoints, if appropriate.
Overall survival | Time from receiving loncastuximab tesirine to death from any cause, assessed at 2 years post-ASCT
  Kaplan-Meier curves and median time-to-event estimation with 95% confidence intervals will be presented for time to-event endpoints, if appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Chow, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No